CLINICAL TRIAL: NCT04681001
Title: Clinical Trial to Evaluate the Efficacy of an Iota-Carrageenan Nasal Spray to Reduce Symptoms Caused by SARS-CoV-2 and Other Respiratory Viruses in Healthcare Workers Managing COVID-19 Patients
Brief Title: Prophylactic Treatment With Carragelose Nasal Spary to Prevent SARS-CoV-2, COVID-19, Infections in Health Care Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVID-19/CHC_20_04
Record Dates: First submitted 2020-12-21; First posted 2020-12-23 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Viral Infection; Common Cold; Severe Acute Respiratory Syndrome (SARS) Pneumonia; COVID-19; Corona Virus Disease
Keywords: Carragelose; Respiratory Virus; Iota-Carrageenan; Health CareWorker; Frontline Worker; Nasal Spray
MeSH Terms: conditions — Common Cold; Severe Acute Respiratory Syndrome; Pneumonia; COVID-19 | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coldamaris pro (Experimental): One puff per nostril three puffs into mouth
  Interventions: Device: nasal spray
- Coldamaris sine (Placebo Comparator): One puff per nostril three puffs into mouth
  Interventions: Device: nasal spray

INTERVENTIONS:
Device: nasal spray — application of nasal spray into nostrils and mouth

SUMMARY:
This is a prospective, randomized placebo-controlled double blinded clinical trial in frontline healthcare workers managing COVID-19 patients. Participants will be weekly tested for SARS-CoV-2 and a panel of respiratory viruses. Treatment will be 3times a day for 84 days one puff into each nostirl and 3 puffs into mouth. Daily a symptom score will be recorded. The primary objective of the trial is to demonstrate that prophylactic treatment of health care workers managing COVID-19 patients with iota-carrageenan reduces symptoms of SARS-CoV-2 infections as well as infections with other respiratory viruses when compared to a placebo-treated control group.

DETAILED DESCRIPTION:
This is a prospective, randomized placebo-controlled double blinded clinical trial in frontline healthcare workers managing COVID-19 patients.

Screening - first day of treatment:

After signing the informed consent form eligible participants will be included. Immediately after inclusion and after first nasal swab, participants start with their first treatment.

In order to obtain nasal swabs and to assess adverse events the participants will visit the sites on a weekly basis over a period of 12 weeks.

3 times a day for 84 days (12 weeks):

* 1 puff of Coldamaris pro. nasal spray into each nostril (1.2 mg/ml; 140 µl per puff) and
* 3 puffs of Coldamaris pro. nasal spray into mouth Weekly sampling for testing of SARS-CoV-2 and respiratory virus panel (Influenza A, Human Metapneumovirus, Influenza A - subtype H1 Adenovirus, Influenza A - subtype H3 Parainfluenza 1, Influenza A - subtype 2009 H1N1, Parainfluenza 2, Influenza B Parainfluenza 3, SARS-CoV-2 Parainfluenza 4, Coronavirus HKU1 Respiratory Syncytial Virus A, Coronavirus N63L, Respiratory Syncytial Virus B, Coronavirus OC43, Rhinovirus/Enterovirus, Coronavirus 229E, Human Bocavirus) At begin and end of trial blood samples will be taken for differential blood count and for serology. The primary end point of the is the presence of COVID-19 symptoms including symptoms of respiratory viral infection. The primary hypothesis is a reduction of symptom days caused by SARS-CoV-2 and/or respiratory viral infection in health care workers treated with Coldamaris pro. nasal spray compared to placebo treated ones

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Study participants that have given informed consent before any study related procedures are performed, and received a copy of signed consent form
* Healthcare workers (nurses, doctors) employed and working at Gesundheitsverbund
* Healthcare workers looking after confirmed COVID-19 positive patients in a secondary care setting such as Accident and Emergency departments, wards, operating theatres, outpatient departments, High Dependency Unit or Intensive Care Units

Exclusion Criteria:

* The subject is related to any study personnel or has any other close ties or conflicts of interest with the study sponsor.
* The subject has received any investigational drug or participated in a clinical trial within 4 weeks of entry to this study
* Known hypersensitivity or allergy to any component of the test product
* Severe cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease or a history or any current disease that is considered by the investigator as a reason for exclusion.
* The subject has a clinically significant disease that could interfere with participation in the study, with the intervention being studied, or with the evaluation of symptoms. Specific exclusions include immune deficiency, autoimmune disease, substantive cardiovascular, endocrinological, neurological, respiratory, or gastrointestinal disease.
* Asymptomatic disease such as elevated blood pressure or cholesterol will not be a reason for exclusion. Those with well-controlled mental illness (e.g. depression, anxiety) will be eligible. The enrolling physician will be empowered to exclude potential subjects that s/he deems unreliable.
* Pregnant women at the time of recruitment will be excluded from the study
* Current medication other than oral contraception, that is considered by the investigator as a reason for exclusion e.g. intranasal medication
* Participation in another antiviral clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Presence of COVID-19 symptoms including symptoms of respiratory viral infection documented in a diary | 84 days
  daily assessment of subjective COVID-19 symptom score

SECONDARY OUTCOMES:
Nasal swabs for analysis of viruses by PCR | 84 days
  weekly assessment of SARS-CoV-2, Influenza A, Human Metapneumovirus, Influenza A - subtype H1, Adenovirus, Influenza A - subtype H3, Parainfluenza 1, Influenza A - subtype 2009 H1N1, Parainfluenza 2, Influenza B, Parainfluenza 3, Parainfluenza 4, Coronavirus HKU1, Respiratory Syncytial Virus A, Coronavirus N63L, Respiratory Syncytial Virus B, Coronavirus OC43, Rhinovirus/Enterovirus, Coronavirus 229E, Human Bocavirus, Chlamydophila pneumoniae, Mycoplasma pneumoniae, Legionella pneumophila
Serology of antibodies against SARS-CoV-2 | 84 days
  beginn and end of trial
Number of viral co-infections dedected by PCR | 84 days
  weekly nasal swabs for analysis of viruses

CONTACTS AND LOCATIONS:
Overall Officials: Iulia Niculescu, MD, Principal Investigator — Gesundheitsverbund; Klinik Favoriten;4. Medizinische Abteilung mit Infektions-und Tropenmedizin1100 Vienna
Locations (2):
- Austria (2):
  - Gesundheitsverbund, Klinik Favoriten, Vienna
  - Gesundheitsverbund Klinik Floridsdorf, Vienna

IPD SHARING:
Plan to Share IPD: No